CLINICAL TRIAL: NCT00129259
Title: Phase II Multiple-Dose Treatment of New Onset Type 1 Diabetes Mellitus With Anti-CD3 mAb
Brief Title: Autoimmunity-blocking Antibody for Tolerance in Recently Diagnosed Type 1 Diabetes
Acronym: AbATE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Immune Tolerance Network (ITN) (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: DAIT ITN027AI
Record Dates: First submitted 2005-08-09; First posted 2005-08-11 (Estimated); Results first posted 2013-09-16 (Estimated); Last update posted 2017-05-22 (Actual); Status verified 2017-04

CONDITIONS: Diabetes Mellitus, Type 1
Keywords: T1D; type 1 diabetes; type 1 diabetes mellitus; juvenile diabetes; autoimmune diabetes; autoimmune; anti-CD3 mAb; mAb hOKT3g1(Ala-Ala); teplizumab
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — teplizumab; ferrous sulfate; Iron-Dextran Complex; FIT1 protein, Arabidopsis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The staff at Northwest Lipid Research Laboratory were masked to the treatment assignment since they performed the mixed-meal tolerance test (MMTT) and the HgA1C assays. All study staff including the PI were masked to the results of the MMTT. They were notified of a detectable or undetectable fasting C-peptide result to assess for continuation to the next treatment cycle.
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Anti-CD3 mAb Plus Diabetes Standard of Care Treatment (Experimental): Subjects receive 1.) a 14-day course of anti-CD3 monoclonal antibody (mAb) intravenously (IV) comprised of daily doses of 51 µg/m2, 103 µg/m2, 207 µg/m2, 413 µg/m2, and 10 days of 826 µg/m2 [Cycle 1] and, when eligible per protocol, receipt of a second 14-day course after a 12-month interval (at month 13)[Cycle 2]. Note: Prior to May 2007, the course of IV daily doses of anti-CD3 mAb were: 57 µg/m2, 115 µg/m2, 230 µg/m2, 460 µg/m2, and 10 days of 919 µg/m2 and, when eligible per protocol, a second course after a 12-month interval (at month 13). 2.) and intensive diabetes standard of care treatment/management under the care of a physician: dietary counseling, insulin dosing and multiple consultations during the course of the trial with the clinical diabetes management team.
  Iron supplementation initiated status post treatment randomization.
  Interventions: Biological: Anti-CD3 mAb; Other: Diabetes Standard of Care Treatment; Dietary Supplement: Iron supplementation
- Diabetes Standard of Care Treatment (Active Comparator): Subjects receive intensive diabetes standard of care treatment/management under the care of a physician: dietary counseling, insulin dosing and multiple consultations during the course of the trial with the clinical diabetes management team.
  Iron supplementation initiated status post treatment randomization.
  Interventions: Other: Diabetes Standard of Care Treatment; Dietary Supplement: Iron supplementation

INTERVENTIONS:
Biological: Anti-CD3 mAb — Daily 14-day dose escalation course at study entry, with possible second course after 12-month interval
  Other Names: mAb hOKT3gamma1(Ala-Ala); teplizumab; MGA031
  Arms: Anti-CD3 mAb Plus Diabetes Standard of Care Treatment
Other: Diabetes Standard of Care Treatment — Receipt of intensive diabetes standard of care treatment/management under the care of a physician: dietary counseling, insulin dosing and multiple consultations during the course of the trial with the clinical diabetes management team.
Dietary Supplement: Iron supplementation — Immediately following randomization, all participants regardless of arm allocation begin iron supplementation with either ferrous sulfate or multivitamin with iron.
  Other Names: MVI; Fer-In-Sol; Feosol; Fer-Iron; Ferolix; FeroSul; Irospan

SUMMARY:
Anti-CD3 monoclonal antibody (a.k.a. hOKT3gamma1 [Ala-Ala],teplizumab, MGA031) is a humanized antibody that is commonly used to prevent organ rejection. The purpose of this study is determine whether anti-CD3 mAb treatment can halt the progression of newly diagnosed type 1 diabetes.

DETAILED DESCRIPTION:
Type 1 diabetes is an autoimmune disease in which the immune system mistakenly attacks insulin-producing beta cells in the pancreas. Without these cells, the body cannot maintain proper blood glucose levels in response to daily activities, such as eating or exercise. Generally, at the time of type 1 diabetes diagnosis, 60% to 85% of the diabetic person's beta cells have already been destroyed. However, between 15% and 40% of these cells remain and are able to produce insulin. Treatment that slows the destruction of additional beta cells may be able to decrease a patient's reliance on insulin and improve their quality of life.

Anti-CD3 mAb is genetically engineered and directed against the CD3 antigen on T cells; this antibody selectively attacks the immune cells responsible for beta cell destruction. In a small exploratory clinical trial, patients with newly diagnosed type 1 diabetes who received a single, 2-week treatment with anti-CD3 mAb had preserved beta cell function and significantly lower insulin requirements than untreated patients for up to two years after therapy. This study will investigate whether a second course of anti-CD3 mAb administered one year after the first administration is able to prolong or improve the effects of the biologic in people who have recently diagnosed type 1 diabetes mellitus.

Participants will be randomly assigned to one of two groups. The Experimental Group will receive anti-CD3 mAb treatment plus Diabetes Standard of Care Treatment; the Active Comparator Group will receive Diabetes Standard of Care Treatment. The Experimental Group will be treated with the antibody for the first 14 days of the study and again one year later. These participants will be admitted to the hospital for the first 5 days of a treatment cycle. Participants who live within 1 hour of the hospital may receive the remainder of a treatment cycle as an outpatient, but those who live farther away will be hospitalized for 14 days. For the first treatment cycle, there will be study visits on the 3 consecutive days after the treatment cycle and at Months 1, 2, 3, 6, 9, and 12. For the second treatment cycle, there will be study visits on the 3 consecutive days after the treatment cycle and at Months 13, 16, 19, 21, and 24.The Active Comparator Group will have 12 study visits over two years.

At study entry, all participants will receive daily iron supplementation, either as ferrous sulfate or a multivitamin with iron. Participants will be followed for up to 2 years to assess their overall diabetes health and to capture laboratory measures of beta cell and immune system function. Medication history and adverse event assessment will occur at all visits. A physical exam, vital signs measurement, and blood collection will occur at most visits. Medical history and urine collection will occur at selected visits.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of type 1 diabetes (according to American Diabetes Association [ADA] criteria) within the 8 weeks prior to study entry
* Weigh at least 25 kg (55 lbs)
* Insulin autoantibodies assessed within 10 days of any insulin use OR anti-glutamic acid decarboxylase (GAD) autoantibodies OR anti-ICA512/IA-2 autoantibodies
* Subjects or guardian(s) willing to provide informed consent

Exclusion Criteria:

* Prior participation in a clinical trial that could potentially affect diabetes condition or immunologic status
* Participation in another investigational clinical trial within the 6 weeks prior to study entry
* Pregnancy or breastfeeding

Ages: 8 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 83 (Actual)
Dates: Start 2005-09; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kevan Herold, MD, Principal Investigator — Yale University
Locations (7):
- United States (7):
  - The Diabetes Center at UCSF, San Francisco, California
  - Barbara Davis Center for Childhood Diabetes, Denver, Colorado
  - Yale University, New Haven, Connecticut
  - Medical College of Georgia, Augusta, Georgia
  - Dept. of Medicine, Division of Endocrinology and the Naomi Berrie Diabetes Center/Columbia University, New York, New York
  - Benaroya Research Institute, Seattle, Washington
  - Pacific Northwest Research Institute/University of Washington, Seattle, Washington

IPD SHARING:
Plan to Share IPD: Yes
Participant level data and additional relevant materials are available to the public in: 1.) the Immunology Database and Analysis Portal (ImmPort), a long-term archive of clinical and mechanistic data from Division of Allergy, Immunology, and Transplantation (DAIT)-funded grants and contracts that also provides data analysis tools available to researchers; and 2.) TrialShare, the Immune Tolerance Network (ITN) Clinical Trials Research Portal that makes data from the consortium's clinical trials publicly available.

REFERENCES:
- [Background] Herold KC, Gitelman SE, Masharani U, Hagopian W, Bisikirska B, Donaldson D, Rother K, Diamond B, Harlan DM, Bluestone JA. A single course of anti-CD3 monoclonal antibody hOKT3gamma1(Ala-Ala) results in improvement in C-peptide responses and clinical parameters for at least 2 years after onset of type 1 diabetes. Diabetes. 2005 Jun;54(6):1763-9. doi: 10.2337/diabetes.54.6.1763. PMID 15919798
- [Background] Herold KC, Hagopian W, Auger JA, Poumian-Ruiz E, Taylor L, Donaldson D, Gitelman SE, Harlan DM, Xu D, Zivin RA, Bluestone JA. Anti-CD3 monoclonal antibody in new-onset type 1 diabetes mellitus. N Engl J Med. 2002 May 30;346(22):1692-8. doi: 10.1056/NEJMoa012864. PMID 12037148
- [Result] Herold KC, Gitelman SE, Ehlers MR, Gottlieb PA, Greenbaum CJ, Hagopian W, Boyle KD, Keyes-Elstein L, Aggarwal S, Phippard D, Sayre PH, McNamara J, Bluestone JA; AbATE Study Team. Teplizumab (anti-CD3 mAb) treatment preserves C-peptide responses in patients with new-onset type 1 diabetes in a randomized controlled trial: metabolic and immunologic features at baseline identify a subgroup of responders. Diabetes. 2013 Nov;62(11):3766-74. doi: 10.2337/db13-0345. Epub 2013 Jul 8. PMID 23835333
- [Derived] Flammer ER, Higdon LE, Sanda S, Garrett TJ, Ismail HM. Baseline Serum Metabolites as Predictors of Teplizumab Response in Individuals with Type 1 Diabetes. medRxiv [Preprint]. 2025 Dec 23:2025.12.22.25342822. doi: 10.64898/2025.12.22.25342822. PMID 41480032
- [Derived] Ajmal N, Bogart MC, Khan P, Max-Harry IM, Healy AM, Nunemaker CS. Identifying Promising Immunomodulators for Type 1 Diabetes (T1D) and Islet Transplantation. J Diabetes Res. 2024 Dec 20;2024:5151171. doi: 10.1155/jdr/5151171. eCollection 2024. PMID 39735417
- [Derived] Boyle KD, Keyes-Elstein L, Ehlers MR, McNamara J, Rigby MR, Gitelman SE, Weiner LJ, Much KL, Herold KC. Two- and Four-Hour Tests Differ in Capture of C-Peptide Responses to a Mixed Meal in Type 1 Diabetes. Diabetes Care. 2016 Jun;39(6):e76-8. doi: 10.2337/dc15-2077. Epub 2016 Apr 13. No abstract available. PMID 27208317
- [Derived] Sherr JL, Ghazi T, Wurtz A, Rink L, Herold KC. Characterization of residual beta cell function in long-standing type 1 diabetes. Diabetes Metab Res Rev. 2014 Feb;30(2):154-62. doi: 10.1002/dmrr.2478. PMID 24115337
- See also: National Institute of Allergy and Infectious Diseases (NIAID) — https://www.niaid.nih.gov/
- See also: Division of Allergy, Immunology, and Transplantation (DAIT) — https://www.niaid.nih.gov/about/dait
- See also: Click here for the Immune Tolerance Network (ITN) TrialShare Web site — https://www.itntrialshare.org/
- See also: Click here for the ITN Website — https://www.immunetolerance.org/
- Available data/document: Individual Participant Data Set: SDY524 — http://www.immport.org/immport-open/public/study/study/displayStudyDetail/SDY524 — ImmPort study identifier is SDY524.
- Available data/document: Study summary, -design (and protocol synopsis), adverse events, medications, demographics, lab tests, study files.: SDY524 — http://www.immport.org/immport-open/public/study/study/displayStudyDetail/SDY524 — ImmPort study identifier is SDY524.
- Available data/document: Individual Participant Data Set: AbaTE - ITN027AI — http://www.itntrialshare.org/project/Studies/ITN027AIDB/Study%20Data/begin.view — TrialShare is the Immune Tolerance Network (ITN) clinical trials research portal that makes data from their clinical trials publicly available without charge.
- Available data/document: Study overview and synopsis, -data and reports, -schedule of assessments, -participant flow diagram, -abstracts and manuscripts: AbaTE-ITN027AI — http://www.itntrialshare.org/project/Studies/ITN027AIDB/Study%20Data/begin.view — TrialShare is the Immune Tolerance Network (ITN) clinical trials research portal that makes data from their clinical trials publicly available without charge.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Seven centers randomized 83 subjects between September 2005 and March 2009. Seventy-seven subjects are in the intent-to-treat (ITT) population. Those not in the ITT population did not have a baseline visit and were not included in the participant flow portion of the results section.
Pre-assignment Details: At a screening visit, subjects underwent procedures to establish that all inclusion criteria were met and none of the exclusion criteria were met. All subjects or guardians provided written informed consent at screening.
Groups:
- Anti-CD3 mAb Plus Diabetes Standard of Care Treatment: Other name: mAb hOKT3gamma1(Ala-Ala), Teplizumab, MGA031. Subjects received 1.) a 14-day course of anti-CD3 monoclonal antibody (mAb) intravenously (IV) comprised of daily doses of 51 µg/m2, 103 µg/m2, 207 µg/m2, 413 µg/m2, and 10 days of 826 µg/m2 [Cycle 1] and, when eligible per protocol, receipt of a second 14-day course after a 12-month interval (at month 13)[Cycle 2]. Note: Prior to May 2007, the course of IV daily doses of anti-CD3 mAb were: 57 µg/m2, 115 µg/m2, 230 µg/m2, 460 µg/m2, and 10 days of 919 µg/m2 and, when eligible per protocol, a second course after a 12-month interval (at month 13). 2.) and intensive diabetes standard of care treatment/management under the care of a physician: dietary counseling, insulin dosing and multiple consultations during the course of the trial with the clinical diabetes management team.
  Iron supplementation was initiated status post treatment randomization.
- Diabetes Standard of Care Treatment: Subjects received intensive diabetes standard of care treatment/management under the care of a physician: dietary counseling, insulin dosing and multiple consultations during the course of the trial with the clinical diabetes management team.
  Iron supplementation was initiated status post treatment randomization.
Period: Overall Study
Arm/Group | Anti-CD3 mAb Plus Diabetes Standard of Care Treatment | Diabetes Standard of Care Treatment
Started | 52 (Subjects not in the Intent-to-treat group did not have a baseline visit and are not included here) | 25 (Subjects not in the Intent-to-treat group did not have a baseline visit and are not included here)
Received All or Part of Cycle 1 | 52 | 0
Received All or Part of Cycle 2 | 40 | 0
Completed | 49 | 22
Not Completed | 3 | 3
Not completed — Lost to Follow-up | 1 | 1
Not completed — Withdrawal by Subject | 2 | 1
Not completed — Only available minimal phone assessments | 0 | 1

BASELINE CHARACTERISTICS:
Population: Intent-to-treat
Groups:
- Anti-CD3 mAb Plus Diabetes Standard of Care Treatment: Other name: mAb hOKT3gamma1(Ala-Ala), Teplizumab, MGA031. Subjects received 1.) a 14-day course of anti-CD3 monoclonal antibody (mAb) intravenously (IV) comprised of daily doses of 51 µg/m2, 103 µg/m2, 207 µg/m2, 413 µg/m2, and 10 days of 826 µg/m2 [Cycle 1] and, when eligible per protocol, receipt of a second 14-day course after a 12-month interval (at month 13)[Cycle 2]. Note: Prior to May 2007, the course of IV daily doses of anti-CD3 mAb were: 57 µg/m2, 115 µg/m2, 230 µg/m2, 460 µg/m2, and 10 days of 919 µg/m2 and, when eligible per protocol, a second course after a 12-month interval (at month 13). 2.) and intensive diabetes standard of care treatment/management under the care of a physician: dietary counseling, insulin dosing and multiple consultations during the course of the trial with the clinical diabetes management team.
- Diabetes Standard of Care Treatment: Subjects received intensive diabetes standard of care treatment/management under the care of a physician: dietary counseling, insulin dosing and multiple consultations during the course of the trial with the clinical diabetes management team.
- Total: Total of all reporting groups
Arm/Group | Anti-CD3 mAb Plus Diabetes Standard of Care Treatment | Diabetes Standard of Care Treatment | Total
Number analyzed (Participants) | 52 | 25 | 77
Age, Continuous [Mean (Standard Deviation); unit: years] | 12.7 (4.9) | 12.3 (4.1) | 12.5 (4.6)
Age, Customized [Number; unit: participants]
  8-12 | 34 | 15 | 49
  13-17 | 14 | 9 | 23
  18-30 | 4 | 1 | 5
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 9 | 33
  Male | 28 | 16 | 44
Region of Enrollment [Number; unit: participants]
  United States | 52 | 25 | 77
C-peptide Area Under the Curve (AUC) Response to a Mixed Meal Tolerance Test (MMTT) at Baseline [Mean (Standard Deviation); unit: pmol/mL] — C-peptide AUC is computed using the trapezoidal rule and dividing by the interval of time from the 4 hour Mixed Meal Tolerance Test (MMTT) where assessments are taken every 30 minutes after initial assessments 15 minutes apart. A higher C-peptide AUC is desirable as detectable C-peptide is a marker for the ability of the pancreas to produce insulin in response to a MMTT.
  pmol/mL | 0.72 (0.29) | 0.67 (0.28) | 0.70 (0.29)
Hemoglobin A1c at Baseline (Pre-treatment) [Mean (Standard Deviation); unit: Percentage (%)] — Glycosylated hemoglobin (HbA1c) is a measure of the average plasma glucose concentration over prolonged periods of time. (Normal :< 5.7%; pre-diabetes: 5.7% -6.4%; diabetes: 6.5% or higher).
  Percentage (%) | 7.4 (0.99) | 7.7 (1.23) | 7.5 (1.07)
Average Total Daily Insulin Dose Per Body Weight at Baseline (Pre-treatment) [Mean (Standard Deviation); unit: Units of Insulin/kilogram/day (U/kg/day)] — This measure is computed using the subject's average amount of exogenous insulin taken per day for the 3 days prior to the visit. (Formula: Total daily insulin dose=total daily insulin requirement (in units of insulin) multiplied by total body weight in kilograms).
  Units of Insulin/kilogram/day (U/kg/day) | 0.39 (0.26) | 0.39 (0.17) | 0.39 (0.23)

OUTCOME MEASURES:

1. Primary Outcome: Change in Mean C-peptide Area Under the Curve (AUC) Response to a Mixed Meal Tolerance Test (MMTT)
Description: C-peptide AUC is computed using the trapezoidal rule and dividing by the interval of time from the 4 hour Mixed Meal Tolerance Test (MMTT) where assessments are taken every 30 minutes after initial assessments 15 minutes apart. A higher C-peptide AUC is desirable as detectable C-peptide is a marker for the ability of the pancreas to produce insulin in response to a MMTT. The baseline data was used to adjust for the C-peptide AUC primary endpoint at 24 months. Missing month 24 C-peptide results are imputed using a conservative scenario.
Time Frame: Baseline (Pre-treatment), Month 24
Population: Intent-to-treat
Measure: Least Squares Mean (95% Confidence Interval); unit: pmol/mL
Arm/Group | Anti-CD3 mAb Plus Diabetes Standard of Care Treatment | Diabetes Standard of Care Treatment
Number analyzed (Participants) | 52 | 25
pmol/mL | -0.28 [-0.36 to -0.20] | -0.46 [-0.57 to -0.35]
Statistical Analysis 1: Comparison: Anti-CD3 mAb Plus Diabetes Standard of Care Treatment vs Diabetes Standard of Care Treatment; Null hypothesis: The mean change from baseline to Month 24 in the 4-hour C-peptide AUC does not differ between treatment groups after adjusting for baseline C-peptide AUC. Alternative hypothesis: The mean change from baseline to Month 24 in the 4-hour C-peptide AUC differs between the treatment groups after adjusting for baseline values; Test type: Superiority or Other; p = 0.002, ANCOVA; P-value for testing treatment effect uses change in ln(AUC+1) as the outcome variable and adjusts for baseline ln(AUC+1)

2. Secondary Outcome: Change in HbA1c
Description: Glycosylated hemoglobin (HbA1c) is a measure of the average plasma glucose concentration over prolonged periods of time and measures the level of optimal management of underlying disease. (Normal :< 5.7%; pre-diabetes: 5.7% -6.4%; diabetes: 6.5% or higher).A decline in HbA1c from baseline to month 24 signifies an improvement in diabetic control. The goal of treatment: to maintain the HgA1c level as close to normal as possible without frequent occurrence of hypoglycemia.
Time Frame: Baseline (Pre-treatment), Month 24
Population: Intent-to-treat with available data
Measure: Mean (Standard Deviation); unit: Percentage (%)
Arm/Group | Anti-CD3 mAb Plus Diabetes Standard of Care Treatment | Diabetes Standard of Care Treatment
Number analyzed (Participants) | 48 | 21
Percentage (%) | 0.129 (2.032) | 0.195 (1.683)
Statistical Analysis 1: Comparison: Anti-CD3 mAb Plus Diabetes Standard of Care Treatment vs Diabetes Standard of Care Treatment; Null hypothesis: The mean change in HbA1c from baseline (pre-treatment) to Month 24 does not differ between treatment groups. Alternative hypothesis: The mean change in HbA1c from baseline to Month 24 differs between treatment groups; Test type: Superiority or Other; p = 0.697, ANCOVA; ANCOVA adjusts for baseline HbA1c

3. Secondary Outcome: Change in Average Total Insulin Dose Per Body Weight
Description: This measure is computed using the average amount of exogenous insulin taken per day for the 3 days prior to the visit. The average insulin use is divided by the subject's weight in kilograms (kg). The need for lower dose(s) of prescribed exogenous insulin while maintaining optimal control of a subject's diabetes reflects improved management of the underlying disease.
Time Frame: Baseline (Pre-treatment), Month 24
Population: Intent-to-treat with available data
Measure: Mean (Standard Deviation); unit: Units of Insulin/kilogram/day (U/kg/day)
Arm/Group | Anti-CD3 mAb Plus Diabetes Standard of Care Treatment | Diabetes Standard of Care Treatment
Number analyzed (Participants) | 46 | 22
Units of Insulin/kilogram/day (U/kg/day) | 0.23 (0.29) | 0.35 (0.28)
Statistical Analysis 1: Comparison: Anti-CD3 mAb Plus Diabetes Standard of Care Treatment vs Diabetes Standard of Care Treatment; Null hypothesis: The mean change from baseline to Month 24 in daily insulin use per kg does not differ between the treatment and control groups. Alternative hypothesis: The mean change from baseline to Month 24 in daily insulin use per kg differs between the treatment and control groups; Test type: Superiority or Other; p = 0.110, ANCOVA; ANCOVA adjusts for baseline daily insulin use per kg

ADVERSE EVENTS:
Time Frame: From the initiation of study treatment through month 24 visit (i.e., throughout the duration of the study)
Description: This study graded the severity of adverse events experienced by the study participant according to criteria set forth in the National Cancer Institute's Common Terminology Criteria for Adverse Events Version 3.0 (June 10, 2003)
Arm/Group | Anti-CD3 mAb Plus Diabetes Standard of Care Treatment | Diabetes Standard of Care Treatment
Serious Adverse Events (participants affected / at risk) | 10/52 | 1/25
Other Adverse Events (participants affected / at risk) | 52/52 | 23/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Anti-CD3 mAb Plus Diabetes Standard of Care Treatment (N=52) | Diabetes Standard of Care Treatment (N=25)
Cytokine release syndrome (Immune system disorders) | 2 (2) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0)
Diarrhoea infectious (Infections and infestations) | 1 (1) | 0 (0)
Infection (Infections and infestations) | 1 (1) | 0 (0)
Skull fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Splenic rupture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Cerebral haemorrhage (Nervous system disorders) | 1 (1) | 0 (0)
Hallucination (Psychiatric disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Anti-CD3 mAb Plus Diabetes Standard of Care Treatment (N=52) | Diabetes Standard of Care Treatment (N=25)
Anaemia (Blood and lymphatic system disorders) | 3 (3) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 12 (24) | 0 (0)
Lymphadenopathy (Blood and lymphatic system disorders) | 4 (4) | 0 (0)
Lymphopenia (Blood and lymphatic system disorders) | 22 (41) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 9 (15) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 5 (5) | 0 (0)
Goitre (Endocrine disorders) | 3 (3) | 1 (1)
Hypothyroidism (Endocrine disorders) | 0 (0) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 16 (20) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 9 (12) | 6 (6)
Constipation (Gastrointestinal disorders) | 5 (6) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 4 (4) | 1 (1)
Nausea (Gastrointestinal disorders) | 25 (43) | 5 (6)
Vomiting (Gastrointestinal disorders) | 19 (34) | 3 (4)
Catheter site rash (General disorders) | 7 (7) | 0 (0)
Chills (General disorders) | 5 (5) | 1 (1)
Fatigue (General disorders) | 7 (9) | 1 (1)
Infusion site pain (General disorders) | 6 (6) | 1 (1)
Malaise (General disorders) | 3 (3) | 2 (2)
Pyrexia (General disorders) | 20 (27) | 5 (5)
Hyperbilirubinaemia (Hepatobiliary disorders) | 3 (4) | 1 (1)
Cytokine release syndrome (Immune system disorders) | 5 (6) | 0 (0)
Seasonal allergy (Immune system disorders) | 3 (3) | 1 (1)
Acne pustular (Infections and infestations) | 5 (6) | 3 (3)
Bronchitis (Infections and infestations) | 3 (3) | 4 (4)
Conjunctivitis infective (Infections and infestations) | 3 (4) | 1 (1)
Diarrhoea infectious (Infections and infestations) | 6 (6) | 2 (2)
Ear infection (Infections and infestations) | 4 (4) | 1 (1)
Gastroenteritis (Infections and infestations) | 3 (3) | 1 (1)
Gastroenteritis viral (Infections and infestations) | 7 (7) | 1 (1)
Influenza (Infections and infestations) | 10 (11) | 5 (8)
Nasopharyngitis (Infections and infestations) | 3 (3) | 1 (1)
Pharyngitis (Infections and infestations) | 11 (14) | 3 (6)
Pharyngitis streptococcal (Infections and infestations) | 1 (1) | 2 (2)
Rhinitis (Infections and infestations) | 5 (6) | 1 (2)
Sinusitis (Infections and infestations) | 5 (5) | 3 (6)
Skin papilloma (Infections and infestations) | 9 (10) | 2 (2)
Tinea infection (Infections and infestations) | 0 (0) | 2 (2)
Upper respiratory tract infection (Infections and infestations) | 32 (80) | 14 (23)
Viral infection (Infections and infestations) | 3 (4) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 5 (5) | 0 (0)
Excoriation (Injury, poisoning and procedural complications) | 8 (12) | 0 (0)
Joint sprain (Injury, poisoning and procedural complications) | 3 (4) | 0 (0)
Alanine aminotransferase increased (Investigations) | 3 (3) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 3 (3) | 0 (0)
CD4 lymphocytes decreased (Investigations) | 5 (5) | 0 (0)
Glycosylated haemoglobin increased (Investigations) | 5 (6) | 8 (8)
Haematocrit decreased (Investigations) | 4 (6) | 0 (0)
Haemoglobin decreased (Investigations) | 7 (10) | 1 (1)
Lymphocyte count decreased (Investigations) | 3 (4) | 0 (0)
Platelet count decreased (Investigations) | 4 (5) | 0 (0)
White blood cell count decreased (Investigations) | 3 (3) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 4 (6) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 21 (26) | 6 (7)
Arthralgia (Musculoskeletal and connective tissue disorders) | 10 (12) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 4 (7) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 7 (12) | 0 (0)
Dizziness (Nervous system disorders) | 8 (9) | 1 (1)
Headache (Nervous system disorders) | 30 (81) | 10 (26)
Tremor (Nervous system disorders) | 5 (7) | 1 (1)
Anxiety (Psychiatric disorders) | 11 (26) | 0 (0)
Ketonuria (Renal and urinary disorders) | 3 (3) | 3 (3)
Dysmenorrhoea (Reproductive system and breast disorders) | 3 (3) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 17 (22) | 3 (4)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3 (5) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 8 (8) | 5 (6)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 12 (19) | 1 (1)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 7 (10) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1)
Tonsillar hypertrophy (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)
Upper respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 4 (6)
Acne (Skin and subcutaneous tissue disorders) | 5 (5) | 1 (1)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 5 (6) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 8 (8) | 1 (1)
Eczema (Skin and subcutaneous tissue disorders) | 3 (5) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 8 (11) | 0 (0)
Lipohypertrophy (Skin and subcutaneous tissue disorders) | 2 (3) | 3 (4)
Pruritus (Skin and subcutaneous tissue disorders) | 15 (25) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 41 (91) | 2 (2)
Rash generalised (Skin and subcutaneous tissue disorders) | 7 (7) | 0 (0)
Rash papular (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0)
Rash pruritic (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0)
Skin exfoliation (Skin and subcutaneous tissue disorders) | 10 (12) | 0 (0)
Hypotension (Vascular disorders) | 12 (18) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No